CLINICAL TRIAL: NCT07151690
Title: A Single-arm Single-center Trial of BCMA/CD3 Bispecific Antibody Treatment for Newly Diagnosed Amyloidosis
Brief Title: BCMA/CD3 Bispecific Antibody Treatment for Newly Diagnosed Amyloidosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025066
Record Dates: First submitted 2025-08-04; First posted 2025-09-03 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-08

CONDITIONS: Systemic Light Chain Amyloidosis
Keywords: Systemic Light Chain Amyloidosis; BCMA/CD3 bispecific antibody; CM336

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BsAbs-treatment group (Experimental): Treatment involves a 12-cycle course of weekly subcutaneous CM336, with step-up dosing during the first week (3 mg on Day 1, 20 mg on Day 4, and 40 mg weekly from Day 8 onward). Dose frequency may be reduced to every two weeks in patients achieving ≥VGPR after 4 cycles.
  Interventions: Drug: anti-BCMA/CD3 bispecific antibody

INTERVENTIONS:
Drug: anti-BCMA/CD3 bispecific antibody — CM336 is a bispecific T-cell engager targeting B-cell maturation antigen (BCMA) and CD3. In this study, CM336 is administered subcutaneously with a step-up dosing strategy in Cycle 1 (3 mg Day 1, 20 mg Day 4, 40 mg Day 8 and onwards weekly). Patients who achieve ≥VGPR by Cycle 4 may switch to 80 mg every two weeks from Cycle 5. The total treatment duration is up to 12 cycles (28 days per cycle), with follow-up for safety and efficacy endpoints including hematologic and organ response.

SUMMARY:
This is a prospective, single-arm, single-center clinical study designed to evaluate the efficacy and safety of low-dose BCMA/CD3 bispecific antibody (CM336) in patients newly diagnosed with systemic light chain (AL) amyloidosis.

ELIGIBILITY:
1. The patient is informed of and voluntarily signs the informed consent form (ICF).
2. Age ≥18 years, regardless of sex.
3. Confirmed diagnosis of primary light-chain (AL) amyloidosis, in accordance with the Guidelines for the Diagnosis and Treatment of Systemic Light-chain Amyloidosis (2021 Revision).
4. Measurable disease at screening, defined as:

   * Difference between involved and uninvolved free light chains (dFLC) ≥50 mg/L, or
   * Serum involved free light chain ≥50 mg/L with an abnormal κ:λ ratio.
5. ECOG performance status ≤2.
6. Adequate organ function within 3 days prior to the first dose of the investigational drug, meeting all of the following criteria:

   i. Absolute neutrophil count (ANC) ≥1.0 × 10⁹/L, with no granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) administration within 7 days, and no pegylated G-CSF administration within 14 days prior to testing; ii. Hemoglobin (Hb) ≥75 g/L, with no whole blood or red blood cell transfusion within 7 days prior to testing; iii. Platelet count ≥70 × 10⁹/L, with no whole blood transfusion, platelet transfusion, or thrombopoietin receptor agonist treatment within 7 days prior to testing; iv. Hepatic function: alanine aminotransferase (ALT) ≤3 × upper limit of normal (ULN), aspartate aminotransferase (AST) ≤3 × ULN, total bilirubin ≤2 × ULN (subjects with Gilbert's syndrome are eligible if direct bilirubin ≤2 × ULN); v. Coagulation: international normalized ratio (INR) or activated partial thromboplastin time (APTT) ≤1.5 × ULN; vi. Renal function: estimated glomerular filtration rate (eGFR) ≥20 mL/min/1.73 m², calculated using the CKD-EPI equation.
7. Male and female patients of childbearing potential, and their partners, must agree to use effective contraceptive methods deemed appropriate by the investigator throughout the treatment period and for at least 3 months thereafter.
8. Male patients must agree not to donate sperm from the screening period until 90 days after the last dose of the investigational drug.
9. The patient must be willing and able to comply with all study procedures and follow-up visits.
10. Women not of childbearing potential are eligible for enrollment. Women of childbearing potential must have a negative serum or urine β-hCG pregnancy test at screening.

Note:

A woman of childbearing potential is defined as a sexually mature woman who has not undergone surgical sterilization (e.g., hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) and has not been postmenopausal for at least 12 consecutive months for reasons other than medical treatment. Women using oral contraceptives or intrauterine devices are considered of childbearing potential. Male subjects (including those who have undergone vasectomy) must agree to use condoms during sexual intercourse with women of childbearing potential and must have no plans to father a child from the time of signing the ICF until 3 months after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Hematologic Very Good Partial Response (VGPR) or Better | From the start of treatment (Day 0), at the end of Cycle 4 (each cycle is 28 days), at the end of Cycle 8 (each cycle is 28 days), and at the end of Cycle 12 (each cycle is 28 days)
  Proportion of participants achieving a hematologic response of VGPR or better (≥VGPR) after 4 treatment cycles of anti-BCMA/CD3 bispecific antibody (CM336), assessed using consensus criteria for AL amyloidosis hematologic response.
Incidence and Severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From the first dose through 30 days after the last dose, up to approximately 24 months.
  Safety will be assessed by monitoring the incidence, nature, and severity of treatment-emergent adverse events (TEAEs), including serious adverse events (SAEs), adverse events of special interest (AESIs) such as cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS), graded according to NCI CTCAE v5.0 and ASTCT criteria. Dose interruptions, modifications, or discontinuations due to toxicity will also be recorded.

SECONDARY OUTCOMES:
Time to First Hematologic Response (TTR) | From the first dose until the best hematologic response (≥PR) is achieved, assessed up to approximately 24 months.
Best Hematologic Response Achieved | From the first dose until the best hematologic response (≥PR) is achieved, assessed up to approximately 24 months.
  The deepest hematologic response (e.g., PR, VGPR, CR, or sCR) observed at any time during the treatment period.
Duration of Hematologic Response (DOR) | From the date of first documented hematologic response to the date of disease progression or death, whichever occurs first, up to approximately 24 months.
  Time from the first documented hematologic response to disease progression or death, whichever occurs first.
Overall Response Rate (ORR) | The overall response rate (ORR) was evaluated at the end of cycle 4, 6, and 12 (28 days per cycle).
Progression-Free Survival (PFS) | From the first dose to progression from any cause, up to approximately 36 months.
Overall Survival (OS) | From the first dose to death from any cause, up to approximately 36 months.
Minimal Residual Disease (MRD) Negativity Rate | At the time of achieving hematologic complete response, up to approximately 24 months.
Standardized uptake value (SUV) | At baseline (prior to first dose), at the end of Cycle 6, and Cycle 12 (each cycle = 28 days)
  Standardized uptake value (SUV) of 18F-92/AV45/TPZA/FT8, 11C-PIB for each target lesion of subject.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided